CLINICAL TRIAL: NCT05983029
Title: Determination of the Utility of the Intergluteal Cleft as a Landmark for nEuraxial Midline identiFication in obsteTric Patients
Brief Title: Determination of Utility of Intergluteal Cleft as Landmark for Neuraxial Midline in Obstetrics
Acronym: CLEFT
Status: Recruiting | Type: Observational
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 291462
Record Dates: First submitted 2022-11-22; First posted 2023-08-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Obstetric Anesthesia Problems

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Each patient will be requested to adopt a standardised upright position. First, two of the investigators will use a spirit level ruler and ink pen to agree upon and visibly mark the horizontal intercristal line on the back of the patient. Second, investigator B will leave the room, and investigator A will make a vertical mark with an ultraviolet pen denoting the intersection of the inferior aspect of the intergluteal cleft and the horizontal intercristal line. Third, investigator A will then leave the room, and investigator B will return to the room to make a vertical mark with an ink pen representing the intersection of the neuraxial midline, as established with the transverse spinous process view on ultrasound, and the horizontal intercristal line. After these two vertical marks have been made at the level of the intercristal line, the horizontal distance between them will be measured in mm by these same two investigators
  Interventions: Diagnostic Test: Intergluteal Cleft; Diagnostic Test: Neuraxial Midline; Diagnostic Test: Horizontal Distance between Vertical Markings

INTERVENTIONS:
Diagnostic Test: Intergluteal Cleft — Marking of intersection between inferior aspect of the intergluteal cleft and the horizontal intercristal line
Diagnostic Test: Neuraxial Midline — Marking of intersection between the neuraxial midline, as established with the transverse spinous process view on ultrasound, and the horizontal intercristal line
Diagnostic Test: Horizontal Distance between Vertical Markings — The horizontal distance between these two vertical marks will be measured at the level of the intercristal line

SUMMARY:
Our aim is to investigate whether a novel landmark, the groove between the buttocks or the intergluteal cleft, can facilitate the identification of the neuraxial midline in obstetric patients when compared to ultrasound as the reference standard for the determination of this midline

DETAILED DESCRIPTION:
Determine if the intergluteal cleft, when compared to ultrasound as the reference standard, can be used to identify the neuraxial midline in obstetric patients

Difference in horizontal distance between the vertical lines of the intergluteal cleft and the neuraxial midline, the latter measured with ultrasound

ELIGIBILITY:
Inclusion criteria

* Female
* 18 years of age or older
* Gestation of 37 weeks or above

Exclusion criteria

* Acute or chronic confusional state
* Allergy to ultrasound gel
* Positive for COVID-19 and/or presence of symptoms consistent with SARS-Cov-2, such as anosmia, cough or fever
* History of previous surgery to the spine
* Scoliosis
* Unable to speak and/or understand English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant patients
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Horizontal distance between intergluteal cleft and neuraxial midline | 12 months
  One horizontal distance and hence one primary outcome

SECONDARY OUTCOMES:
Difference in horizontal distance stratified by body mass index | 12 months
  Variation for BMI and recorded data
Difference in horizontal distance stratified by presence of pre-eclampsia | 12 months
  Variation for pre-ecalmpsia and recorded data
Difference in horizontal distance stratified by presence of pregnancy induced hypertension | 12 months
  Variation for pregnancy induced hypertension a and recorded data

CONTACTS AND LOCATIONS:
Overall Officials: Gill Arbane, BSc, Study Chair — Guys' & St Thomas' NHS Foundation Trust
Locations (1):
- Guy's Hospital, Great Maze Pond, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No